CLINICAL TRIAL: NCT06402955
Title: Identifying the Neural Basis of Depression in Parkinson's Disease
Brief Title: Imaging Depression in Parkinson's Disease
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Principal Investigator, Sophie Holmes, Assistant Professor of Psychiatry, Yale University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2000037090; R01NS125482-01A1 (NIH)
Record Dates: First submitted 2024-05-02; First posted 2024-05-07 (Actual); Last update posted 2025-07-14 (Actual); Status verified 2025-07

CONDITIONS: Parkinson's Disease; Major Depressive Disorder
Keywords: Imaging
MeSH Terms: conditions — Parkinson Disease; Depressive Disorder, Major | interventions — 1-((3-(methylpyridin-4-yl)methyl)-4-(3,4,5-trifluorophenyl)pyrrolidin-2-one; Ketamine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Parkinson's Disease with Major Depressive Disorder (Other): This study aims to identify mechanisms unique to patients with both Parkinson's Disease and Major Depressive Disorder.
  Interventions: Radiation: 11C-UCB-J; Drug: ketamine hydrochloride

INTERVENTIONS:
Radiation: 11C-UCB-J — Radiotracer for imaging
Drug: ketamine hydrochloride — There will be a small subset (opt-in) who will receive a single dose of ketamine to determine the ability of ketamine to target these mechanisms and initiate an associated antidepressant response. If the participant is opting into the ketamine arm, the investigators will ask them to come in for one single-dose of ketamine and complete another PET and MRI scan post-ketamine treatment.

SUMMARY:
The goal of this observational study is to identify targetable neural substrates of depression in Parkinson's Disease for the first time in people with Parkinson's between the ages of 40 and 80, who are experiencing symptoms of depression.

DETAILED DESCRIPTION:
This study will compare people with Parkinson's Disease and depression to individuals with Parkinson's Disease without Major Depressive Disorder, Major Depressive Disorder with no Parkinson's, and Healthy Controls. Up to 30 participants will be recruited and enrolled for each of these 4 groups. Participants will be asked to complete one PET and one MRI scan along with study assessments. Once screening and consent is completed, participants will be scheduled for PET and MRI scans. The total duration for participants in this study is 7 hours, including the screening visit and then one additional visit for the scans.

There will also be a small subset (opt-in) who will receive a single dose of ketamine to determine the ability of ketamine to target these mechanisms and initiate an associated antidepressant response. If the participant is opting into the ketamine arm, the investigators will ask them to come in for one single-dose of ketamine and complete another PET and MRI scan post-ketamine treatment.

The main questions it aims to answer are: 1) Will the Parkinson's depression group exhibit a distinct pattern of synaptic deficits compared to other groups? 2) Will there be differences in functional connectivity across groups? 3) Are there associations between synaptic density and functional connectivity across groups? 4) Will ketamine increase synaptic density in PD-affected and mood-related circuitry, and will that be associated with an antidepressant response?

ELIGIBILITY:
Inclusion Criteria:

1. Age 40-80.
2. For women of reproductive potential, a negative pregnancy test at screening and scanning
3. For PD patients, clinical diagnosis of PD, able to consent and tolerate PET procedures
4. For PD depression patients - at least moderate symptom severity as determined by at least 15 on the MADRS, which has shown maximum discrimination between depressed and non-depressed PD patients.
5. For dPD patients undergoing ketamine, abstinence from drugs of abuse, other than alcohol, cannabis, nicotine and caffeine for the duration of the study. Patients with substance use disorders as defined by the DSM-5 will be excluded.

Exclusion Criteria:

1. Dementia (Montreal Cognitive Assessment (MoCA) score <21)
2. A significant primary DSM-5 psychiatric disorder except for MDD
3. A history of or current significant medical (e.g. cardiovascular, renal), or neurological (e.g. cerebrovascular, seizure, traumatic brain injury) illness other than PD that is unstable and significantly increase their risk and/or might affect the study objectives, as determined by study physicians.
4. Prior radiation exposure for research purposes within such that participation in this study would place them over FDA limits for annual radiation exposure
5. Medications affecting SV2A availability (e.g. levetiracetam)
6. For dPD patients receiving ketamine, uncontrolled hypertension, defined as average blood pressure greater than or equal to 140 mmHg or an average diastolic blood pressure greater than or equal to 90 mmHg among those patients who have hypertension.
7. Contraindications to MRI.
8. For patients undergoing arterial sampling for the PET scan: Iodine allergy, bleeding disorder and/or use of blood thinning medication
9. Inability to provide written informed consent according to the Yale Human Investigation Committee (HIC) guidelines in English.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2025-12-01 (Estimated); Primary Completion 2029-04 (Estimated); Study Completion 2029-12 (Estimated)

PRIMARY OUTCOMES:
Montgomery-Åsberg Depression Rating Scale (MADRS) | One day
  This assessment stratifies severity of depressive episodes in adults. Ratings are based on clinical interview with the patient. Use clinical judgment to determine whether the rating lies on the defined scale steps (0, 2, 4, 6 points) or between them (1, 3, 5 points, denoted as "(Worsening symptoms)").The MADRS scoring instructions indicate that a total score ranging from 0 to 6 indicates that the patient is in the normal range (no depression), a score ranging from 7 to 19 indicates "mild depression," 20 to 34 indicates "moderate depression," a score of 35 and greater indicates "severe depression," and a total score of 60 or greater indicates "very severe depression."

SECONDARY OUTCOMES:
Binding potential (BPND) | One week
  Binding potential (BPND) reflects the ratio at equilibrium of specifically bound radioligand to that of non-displaceable radioligand in tissue. BPND maps will be generated using the simplified reference tissue method 2 (SRTM2) and the centrum semiovale (CS) as reference region.

CONTACTS AND LOCATIONS:
Locations (1):
- Yale University, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: Undecided